CLINICAL TRIAL: NCT06456528
Title: Phase 2/3 Randomized, Double-blind, Placebo-controlled Study of QL0911 for the Treatment of Cancer Treatment-Induced Thrombocytopenia.
Brief Title: QL0911 for the Treatment of Cancer Treatment-Induced Thrombocytopenia
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QL0911-302
Record Dates: First submitted 2024-06-07; First posted 2024-06-13 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Cancer Treatment-Induced Thrombocytopenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- QL0911 (Experimental)
  Interventions: Drug: QL0911
- QL0911 plus Placebo (Experimental)
  Interventions: Drug: QL0911 plus Placebo
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: QL0911 — QL0911
  Arms: QL0911
Drug: QL0911 plus Placebo — QL0911 plus Placebo
  Arms: QL0911 plus Placebo
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
To evaluate the efficacy and safety of QL0911 in cancer treatment-induced thrombocytopenia. Thrombocytopenia is a low number of platelets in the blood. Sometimes, thrombocytopenia is a side effect of cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, 18-75 years of age;
* Histopathological or cytological examination confirmed cancer , chemotherapy cycle of 21 days;
* Participant experienced thrombocytopenia and chemotherapy delay;
* ECOG performance status 0-1;
* The estimated survival time at screening is ≥12 weeks, and the current chemotherapy regimen can be accepted for at least 2 cycles.

Exclusion Criteria:

* Participant has any history of hematologic diseases other than chemotherapy-induced thrombocytopenia;
* Participant has serious bleeding symptoms;
* History of allergy to the study drug;
* Patients with hepatitis C antibody positive and detection of HCV-RNA exceeding the upper limit, patients with hepatitis B surface antigen positive and detection of HBV-DNA exceeding the upper limit, patients with severe cirrhosis, HIV antibody positive and syphilis antibody positive;
* Pregnant or lactating women;
* Participant has received any experimental therapy within 28 days prior to screening
* Other conditions that may affect participant's safety or trial evaluations per investigator's discretion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The proportion of treatment responders. | Randomization up to 80 days

SECONDARY OUTCOMES:
Duration from the commencement of treatment to a platelet count ≥100×109/L | Randomization up to 30 days
Proportion of subjects who could complete chemotherapy without dose modification and rescue therapy | Randomization up to 150 days
Number of adverse events (AEs)/serious adverse events (SAEs) | Randomization up to 150 days

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Harbin First Hospital, Harbin
  - Nanjing Tianyinshan Hospital, Nanjing